CLINICAL TRIAL: NCT00981799
Title: A Phase I Trial of NECTAR (Nelarabine, Etoposide and Cyclophosphamide in T-ALL Relapse): A Joint Study of TACL and POETIC
Brief Title: Trial of Nelarabine, Etoposide and Cyclophosphamide in Relapsed T-cell ALL and T-cell LL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual rate
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2008-002
Record Dates: First submitted 2009-09-09; First posted 2009-09-22 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Relapsed T-Cell Acute Lymphoblastic Leukemia; Relapsed T-Cell Lymphoblastic Lymphoma
Keywords: Relapse; T cell; Lymphoblastic; Leukemia; Lymphoma; Nelarabine; TACL; NECTAR
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Leukemia; Lymphoma | interventions — nelarabine; Etoposide; etoposide phosphate; Cyclophosphamide; Methotrexate; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nelarabine Dose Level 1 (Experimental): The study will begin at Dose Level 1 at 480 mg/m2 Nelarabine (75% of single agent maximum tolerated dose) and 330 mg/m2 Cyclophospamide and will escalate to the next Dose Level if the maximum tolerated dose (MTD) is not exceeded. The first 3 patients will be enrolled into Dose Level 1. If 0/3 experiences dose limiting toxicity (DLT) at a given dose level, then the dose is escalated to the next higher level and 3 more patients are enrolled. If 1/3 experiences DLT at current dose, the up to 3 more patients are accrued at the same dose level. If 2 or more DLTs are observed in a 3-patient or 6-patient cohort at a given dose level, then the MTD has been exceeded, dose escalation will be stopped, and up to 3 additional patients will be enrolled at the next lower dose level (unless 6 patients have already been treated at that prior dose). If the MTD is exceeded at Dose Level 0, the study will be closed.
  Interventions: Drug: Nelarabine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Filgrastim
- Nelarabine Dose Level 2 (Experimental): Patients in this arm will be administered Nelarabine at 650 mg/m2 (100% of single agent MTD) and 330 mg/m2 Cyclophosphamide.
  Interventions: Drug: Nelarabine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Filgrastim
- Nelarabine Dose Level 3 (Experimental): Patients in this arm will be administered Nelarabine at 650 mg/m2 (100% of single agent MTD) and 400 mg/m2 Cyclophosphamide
  Interventions: Drug: Nelarabine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Filgrastim
- Nelarabine Dose Level 0 (Experimental): Patients in this arm will be administered Nelarabine 325 mg/m2 (50% of single agent MTD) and 330 mg/2 Cyclophosphamide. Patients will only enter this arm if the MTD at Dose Level 1 has been exceeded. If the MTD is exceeded at Dose Level 0, the study will be closed.
  Interventions: Drug: Nelarabine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Filgrastim

INTERVENTIONS:
Drug: Nelarabine — Dose will be assigned at study entry. Nelarabine will be given IV over 60 minutes (given at hours 0 to 1) on days 1 through 5.
  Other Names: Arranon; Compound 506U78
Drug: Etoposide — 100 mg/m2/day IV over 2 hours (given at hours 1 to 3) on days 1 through 5
  Other Names: VePesid; Etopophos; VP-16
Drug: Cyclophosphamide — Dose will be assigned at study entry, IV as a 30-60 minute infusion (given at hours 3 to 4) on days 1 through 5.
  Other Names: Cytoxan
Drug: Methotrexate — Give between day 29 and 36 or when ANC>750 and PLTS>75,000 - whichever comes first (but not prior to day 22) at the dose defined by age below, ideally in conjunction with BM evaluation.
  Given intrathecally at the dose defined by age below. 8 mg for patients age greater than or equal to 1, but <2 years of age 10 mg for patients age greater than or equal to 2, but <3 years of age 12 mg for patients greater than or equal to 3, but < 9 years of age 15 mg for patients greater than or equal to >9 years of age
  Other Names: MTX; Amethopterin; Trexall
Drug: Filgrastim — 5 micrograms/kg/day IV or SC will begin on Day 6 and end when the ANC is > 1000/mm3 for two consecutive days.
  Other Names: Neupogen; GCSF; granulocyte colony stimulating factor

SUMMARY:
Nelarabine has shown significant activity in patients with T-cell malignancies. This study will determine the safety and maximum tolerated dose of the combination of nelarabine, cyclophosphamide and etoposide in patients with first bone marrow relapse of T-ALL, or first relapse of T-LL.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be enrolled in the dose-escalation portion of this study must have T-cell ALL or T-cell lymphoblastic lymphoma (LL) in first relapse or must have failed primary induction chemotherapy (ie, never attained a complete remission following an initial course of standard therapy for T-ALL or T-LL). Patients to be enrolled in the cohort expansion portion of this study (ie, those treated at the recommended phase 2 dose) must have T-cell ALL in first relapse or must have failed primary induction chemotherapy (ie, never attained a complete remission following an initial course of standard therapy for T-ALL). T-LL patients are not eligible for the cohort expansion phase.
* Patients with T-cell ALL must have greater than 25% blasts in the bone marrow with or without extramedullary disease.
* Patients with T-cell LL must have recurrent disease, documented by clinical or radiographic criteria, as well as histologic verification of the malignancy at original diagnosis. Patients with T-cell LL enrolled in the phase I dose-escalation study are not required to have measurable disease; however, patients enrolled in the phase II cohort expansion at the MTD must have measurable disease.
* Patients may have CNS 1 or CNS 2 disease but not CNS 3.
* ECOG 0-2 or Karnofsky ≥ 50% for patients > 16 years of age; Lansky ≥ 50% for patients ≤16 years of age.
* Patients may be enrolled on study regardless of the timing of prior Intrathecal therapy; however, they MAY NOT BEGIN TREATMENT ON THIS PROTOCOL UNTIL A MINIMUM OF 7 DAYS HAS ELAPSED SINCE PRIOR INTRATHECAL THERAPY.
* At least 6 weeks must have elapsed since administration of nitrosureas.
* At least 12 weeks must have elapsed since administration of craniospinal or hemipelvic radiation.
* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.
* Adequate renal function defined as serum creatinine ≤ 1.5x upper limit of normal (ULN) for age. If the serum creatinine is above these values, the calculated creatinine clearance or radioisotope GFR must be ≥ 70 mL/min/1.73m2.
* Total bilirubin ≤ 1.5x ULN for age. If the total bilirubin is elevated, patient will still be eligible if the conjugated (direct) serum bilirubin ≤ ULN for age.
* ALT ≤ 5x ULN of normal for age.
* Adequate cardiac function defined as shortening fraction of ≥ 27% by echocardiogram or ejection fraction ≥ 45% by gated radionuclide study.
* No evidence of dyspnea at rest
* No exercise intolerance
* A pulse oximetry ≥ 94% at sea level (≥ 90% at altitude ≥ 5000 feet) if there is clinical indication for determination.
* Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

* Patients with Down syndrome are excluded.
* Patients with pre-existing Grade 2 (or greater) peripheral motor or sensory neurotoxicity per the CTCAE 3.0 as determined by the treating physician or a neurologist.
* Patients with a history of prior veno-occlusive disease (VOD) or findings consistent with a diagnosis of VOD, defined as: conjugated serum bilirubin >1.4 mg/dL AND unexplained weight gain greater than 10% of baseline weight or ascites AND hepatomegaly or right upper quadrant pain without another explanation, OR reversal of portal vein flow on ultrasound, OR pathological confirmation of VOD on liver biopsy.
* Previous hematopoetic stem cell transplantation.
* Patients with a prior seizure disorder requiring anti-convulsant therapy are not eligible to receive nelarabine. For the purposes of this study, this includes any patient that has received anticonvulsant therapy to prevent/treat seizures in the prior two years.
* Positive blood culture within 48 hours of study enrollment.
* Fever above 38.2 within 48 hours of study enrollment with clinical signs of infection.
* Plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-06; Primary Completion 2015-11 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Whitlock, MD, Study Chair — The Hospital for Sick Children
Locations (37):
- United States (26):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - New York University Medical Center, New York, New York
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Rainbow Babies, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Jude, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas at Southwestern, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Primary Children's, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Melbourne, Victoria
  - Sydney Children's Hospital, Sydney
- St. Anna Children's Hospital, Vienna, Austria
- Canada (3):
  - Hospital for Sick Kids, Toronto, Ontario
  - Sainte Justine University Hospital, Montreal, Quebec
  - British Columbia Children's Hospital, Vancouver
- CHU Lille, Lille, France
- Bambino Gesù Hospital, Rome, Italy
- Erasmus MC - Sophia, Rotterdam, Netherlands

REFERENCES:
- See also: For more information about this and other clinical trials, please visit the TACL website — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Nelarabine Dose Level 1: The study will begin at Dose Level 1 at 480 mg/m2 Nelarabine (75% of single agent maximum tolerated dose) and 330 mg/m2 Cyclophospamide and will escalate to the next Dose Level if the maximum tolerated dose (MTD) is not exceeded.
  Nelarabine: Dose will be assigned at study entry. Nelarabine will be given IV over
- Nelarabine Dose Level 0: Patients in this arm will be administered Nelarabine 325 mg/m2 (50% of single agent MTD) and 330 mg/2 Cyclophosphamide. Patients will only enter this arm if the MTD at Dose Level 1 has been exceeded. If the MTD is exceeded at Dose Level 0, the study will be closed.
  Nelarabine: Dose will be assigned at study entry. Nelarabine will be given IV over 60 minutes (given at hours 0 to 1) on days 1 through 5.
  Etoposide: 100 mg/m2/day IV over 2 hours (given at hours 1 to 3) on days 1 through 5
  Cyclophosphamide: Dose will be assigned at study entry, IV as a 30-60 minute infusion (given at hours 3 to 4) on days 1 through 5.
  Methotrexate: Give between day 29 and 36 or when ANC>750 and PLTS>75,000 - whichever comes first (but not prior to day 22) at the dose defined by age below, ideally in conjunction with BM evaluation.
  Given intrathecally at the dose defined by age below. 8 mg for patients age greater than or equal to 1, but <2 years of age 10 mg for patients age greater than
Period: Overall Study
Arm/Group | Nelarabine Dose Level 1 | Nelarabine Dose Level 2 | Nelarabine Dose Level 3 | Nelarabine Dose Level 0
Started | 6 | 7 | 10 | 0
Completed | 5 | 6 | 10 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dose Level 0 did not accrue any subjects as the criteria to accrue at Dose Level 0 was not met
Groups:
- Nelarabine Dose Level 1: The study will begin at Dose Level 1 at 480 mg/m2 Nelarabine (75% of single agent MTD) and 330 mg/m2 Cyclophosphamide. The first 3 patients will be enrolled into Dose Level 1.
  If 0/3 experiences dose limiting toxicity (DLT) at a given dose level, then the dose is escalated to the next higher level and 3 more patients are enrolled. If 1/3 experiences DLT at current dose, the up to 3 more patients are accrued at the same dose level. If 2 or more DLTs are observed in a 3-patient or 6-patient cohort at a given dose level, then the MTD has been exceeded, dose escalation will be stopped, and up to 3 additional patients will be enrolled at the next lower dose level (unless 6 patients have already been treated at that prior dose). If the MTD is exceeded at Dose Level 0, the study will be closed.
- Nelarabine Dose Level 2: Patients in this arm will be administered Nelarabine at 650 mg/m2 (100% of single agent MTD) and 330 mg/m2 Cyclophosphamide.
  This is the second dose level of this dose escalation study. If 1 or fewer patients at Dose Level 1 experiences a DLT, patients will be accrued at Dose Level 2.
  If 0/3 experiences dose limiting toxicity (DLT) at a given dose level, then the dose is escalated to the next higher level and 3 more patients are enrolled. If 1/3 experiences DLT at current dose, the up to 3 more patients are accrued at the same dose level. If 2 or more DLTs are observed in a 3-patient or 6-patient cohort at a given dose level, then the MTD has been exceeded, dose escalation will be stopped, and up to 3 additional patients will be enrolled at the next lower dose level (unless 6 patients have already been treated at that prior dose). If the MTD is exceeded at Dose Level 0, the study will be closed.
- Nelarabine Dose Level 3: Patients in this arm will be administered Nelarabine at 650 mg/m2 (100% of single agent MTD) and 400 mg/m2 Cyclophosphamide This is the third and final dose level of this dose escalation study. If 1 or fewer patients at Dose Level 2 experiences a DLT, patients will be accrued at Dose Level 3.
  If 0/3 experiences dose limiting toxicity (DLT) at a given dose level, then the dose is escalated to the next higher level and 3 more patients are enrolled. If 1/3 experiences DLT at current dose, the up to 3 more patients are accrued at the same dose level. If 2 or more DLTs are observed in a 3-patient or 6-patient cohort at a given dose level, then the MTD has been exceeded, dose escalation will be stopped, and up to 3 additional patients will be enrolled at the next lower dose level (unless 6 patients have already been treated at that prior dose). If the MTD is exceeded at Dose Level 0, the study will be closed.
- Total: Total of all reporting groups
Arm/Group | Nelarabine Dose Level 1 | Nelarabine Dose Level 2 | Nelarabine Dose Level 3 | Nelarabine Dose Level 0 | Total
Number analyzed (Participants) | 6 | 7 | 10 | 0 | 23
Age, Continuous [Mean (Full Range); unit: years] | 13 [9 to 18] | 7 [1 to 15] | 10.5 [5 to 17] |  | 9 [1 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 0 | 8
  Male | 4 | 4 | 7 | 0 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 |  | 2
  Not Hispanic or Latino | 4 | 6 | 9 |  | 19
  Unknown or Not Reported | 1 | 0 | 1 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 1 | 2 | 4 |  | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 |  | 1
  Black or African American | 1 | 0 | 3 |  | 4
  White | 3 | 4 | 3 |  | 10
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 0 | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Presence of Dose-limiting Toxicities (DLTs) of Nelarabine, Etoposide and Cyclophosphamide When Given in Combination to Children With T-ALL and Bone Marrow Relapse or T-LL.
Description: Patients will be evaluated based on Dose Level and total courses taken at each dose level and for presence of dose limiting toxicities. Not all patients enrolled at each dose level has been assessed to be evaluable for DLTs. Only those that have met criteria for being evaluable for DLT will be counted in the Overall Number of Participants Analyzed.
Time Frame: 6 months
Population: There are 0 patients for Dose Level 0 as no patients met the criteria to be enrolled
Measure: Count of Participants; unit: Participants
Groups:
- Nelarabine Dose Level 1: The study will begin at Dose Level 1 at 480 mg/m2 Nelarabine (75% of single agent maximum tolerated dose) and 330 mg/m2 Cyclophospamide and will escalate to the next Dose Level if the maximum tolerated dose (MTD) is not exceeded.
Arm/Group | Nelarabine Dose Level 1 | Nelarabine Dose Level 2 | Nelarabine Dose Level 3 | Nelarabine Dose Level 0
Number analyzed (Participants) | 5 | 6 | 10 | 0
Participants
  # of patients with DLT | 0 | 1 | 2 | 0
  # of patients without DLT | 5 | 5 | 8 | 0

2. Secondary Outcome: To Determine the Complete Remission Rate After 1 and 2 Courses of This Therapy in Children With T-ALL and Bone Marrow Relapse or T-LL.
Description: Patients will be evaluated at each dose level and for assessment of response to treatment. Not all patients enrolled at each dose level has been assessed to be evaluable for response. Only those that have met criteria for being evaluable for response will be counted in the Overall Number of Participants Analyzed.
Time Frame: 1-3 months
Population: No patients met the criteria to be enrolled at Dose Level 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Nelarabine Dose Level 1 | Nelarabine Dose Level 2 | Nelarabine Dose Level 3 | Nelarabine Dose Level 0
Number analyzed (Participants) | 5 | 6 | 10 | 0
Participants
  # of patients not with complete remission | 3 | 4 | 9 | 0
  # of patients with complete remission | 2 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose of Nelarabine, Etoposide, and Cyclophosphamide until 30 days following the last dose of protocol therapy (approximately from Day 0 to Day 66)
Description: The definitions of AE and SAE do not differ from the clinicaltrials.gov definitions
Groups:
- Nelarabine Dose Level 1: The study will begin at Dose Level 1 at 480 mg/m2 Nelarabine (75% of single agent maximum tolerated dose) and 330 mg/m2 Cyclophospamide and will escalate to the next Dose Level if the maximum tolerated dose (MTD) is not exceeded. The first 3 patients will be enrolled into Dose Level 1.
Arm/Group | Nelarabine Dose Level 1 | Nelarabine Dose Level 2 | Nelarabine Dose Level 3 | Nelarabine Dose Level 0
All-Cause Mortality (participants affected / at risk) | 4/6 | 7/7 | 8/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 5/7 | 7/10 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 10/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelarabine Dose Level 1 (N=6) | Nelarabine Dose Level 2 (N=7) | Nelarabine Dose Level 3 (N=10) | Nelarabine Dose Level 0 (N=0)
HLH-Syndrome-Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0
Neuropathy- Peripheral Motor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0
Neuropathy- Peripheral Sensory (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0
Infection, Parainfluenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0
Herpes Zoster Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0
Oral Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0
Infection Oral cavity (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4) | 0
Infection, vulva (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0
Infection, perianal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0
catheter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Hypoalbuminemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0
hyponatremia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0
elevated bilirubin (Investigations) | 0 | 1 (1) | 0 | 0
GI bleed (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Sepsis (Immune system disorders) | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelarabine Dose Level 1 (N=6) | Nelarabine Dose Level 2 (N=7) | Nelarabine Dose Level 3 (N=10) | Nelarabine Dose Level 0 (N=0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (4) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Epistaxis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (3) | NA
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 10 (10) | NA
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | NA
Hypocalcemia (Investigations) | 3 (3) | 1 (1) | 1 (1) | NA
Hypokalemia (Investigations) | 3 (3) | 2 (2) | 3 (3) | NA
Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | NA
Leukopenia NOS (Blood and lymphatic system disorders) | 3 (3) | 5 (6) | 5 (5) | NA
Muscle weakness, lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Neutrophil count (Investigations) | 1 (1) | 6 (7) | 4 (4) | NA
Pain NOS (General disorders) | 1 (1) | 0 (0) | 1 (1) | NA
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | NA
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | NA
Hyperuricemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 6 (8) | NA
Anorexia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | NA
aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | NA
blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
clostridial infection NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
constitutional symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | NA
diarrhea NOS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | NA
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Hyperkalemia (Investigations) | 0 (0) | 2 (2) | 0 (0) | NA
Hypernatremia (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
Hyponatremia (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
hypoxia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | NA
Infection, blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Influenza like illness (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
lymphopenia (Endocrine disorders) | 0 (0) | 4 (5) | 6 (6) | NA
metabolic lab -other (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
nausea (General disorders) | 0 (0) | 2 (2) | 1 (1) | NA
Pain other (General disorders) | 0 (0) | 1 (1) | 1 (1) | NA
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | NA
Platelet count decrease (Blood and lymphatic system disorders) | 0 (0) | 6 (8) | 10 (11) | NA
pulmonary hypertension NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Pyrexia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
vomiting (General disorders) | 0 (0) | 1 (1) | 1 (1) | NA
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Allergy/Immunology- Other (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Catheter-related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days